CLINICAL TRIAL: NCT04863976
Title: Effects of Different Stretching Techniques on Extensibility, Strength and Range of Motion in Football Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Luis Ceballos Laita, Ph.D, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI21 - 2213
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Asymptomatic Condition
Keywords: stretching; extensibility; strength; range of motion
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic stretching (Experimental)
  Interventions: Other: Dynamic stretching
- Passive stretching (Active Comparator)
  Interventions: Other: Passive stretching
- Self-stretching (Active Comparator)
  Interventions: Other: Self-stretching

INTERVENTIONS:
Other: Dynamic stretching — Dynamic movements of the joints controlled by the quadriceps muscle (hip and knee)
  Arms: Dynamic stretching
Other: Passive stretching — passive stretching of the quadriceps muscle
  Arms: Passive stretching
Other: Self-stretching — Self-stretching of the quadriceps muscle
  Arms: Self-stretching

SUMMARY:
To compare the effects dynamic stretching, passive stretching and self-stretching of the quadriceps muscle on muscle extensibility, hip strength and hip range of motion

ELIGIBILITY:
Inclusion Criteria:

* Footbal athletes
* Limited range of motion in ely's test

Exclusion Criteria:

* Previous surgery in the lower limb
* Previous physiotherapy threatment in the thigh
* Stretching contraindications

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Range of motion | Baseline
  the examiners assess the shoulder range of motion with an universal goniometer
  the examiners assess the shoulder range of motion with an universal goniometer
  The examiners assess the hip flexion and extension range of motion with an universal goniometer
Range of motion | immediately after the intervention
  the examiners assess the shoulder range of motion with an universal goniometer
  the examiners assess the shoulder range of motion with an universal goniometer
  The examiners assess the hip flexion and extension range of motion with an universal goniometer
Strength | Baseline
  The examiners assess the hip flexion and extension strength with a hand-held dynamometer
Strength | immediately after the intervention
  The examiners assess the hip flexion and extension strength with a hand-held dynamometer
Extensibility | Baseline
  The examiners assess the extensibility of the quadriceps and hamstring tissues using a digital inclinometer
Extensibility | immediately after the intervention
  The examiners assess the extensibility of the quadriceps and hamstring tissues using a digital inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ceballos Laita, PhD, Principal Investigator — University of Valladolid
Locations (1):
- Luis Ceballos Laita, Soria, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No